CLINICAL TRIAL: NCT00660699
Title: A Feasibility Phase II Study of Gemcitabine With Docetaxel With Concurrent 3-D Conformal Radiation Plus Continuous Infusion 5-Fluorouracil in the Treatment of Resected Cholangiocarcinoma, Gallbladder, Pancreatic and Ampullary Cancers
Brief Title: A Feasibility Phase II Study in the Treatment of Resected Cholangiocarcinoma, Gallbladder, Pancreatic and Ampullary Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-0580 / 201101866
Record Dates: First submitted 2008-04-11; First posted 2008-04-17 (Estimated); Results first posted 2015-05-27 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Cholangiocarcinoma Cancer; Gallbladder Cancer; Pancreatic Cancer; Ampullary Cancer
Keywords: Cholangiocarcinoma; Gallbladder; Pancreatic; Ampullary; Cancer
MeSH Terms: conditions — Gallbladder Neoplasms; Pancreatic Neoplasms; Cholangiocarcinoma; Neoplasms | interventions — Gemcitabine; Docetaxel; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (gemcitabine, docetaxel, 5FU, radiation) (Experimental): Gemcitabine 1000 mg/m2 IV on Day 1 and Day 8 of a 21 day cycle for 2 cycles
  Docetaxel 35 mg/m2 IV on Day 1 and Day 8 of a 21 day cycle for 2 cycles
  5FU CIVI 225 mg/m2 per day throughout radiation (starts 3 weeks after start of cycle 2)
  Radiation 5040 cGy or 5400 cGy for positive margins (starts 3 weeks after start of cycle 2). Daily dose of 1.8 Gy five days per week.
  Gemcitabine 1000 mg/m2 IV on Days 1 and 8 of 21 day cycle for 2 cycles (this starts 4 weeks after radiation)
  Docetaxel 35 mg/m2 IV on Days 1 and 8 of 21 day cycle for 2 cycles (this starts 4 weeks after radiation)
  Interventions: Drug: Gemcitabine; Drug: Docetaxel; Radiation: Radiation

INTERVENTIONS:
Drug: Gemcitabine
  Other Names: Gemzar
Drug: Docetaxel
  Other Names: Taxotere
Radiation: Radiation

SUMMARY:
To assess the feasibility of administering induction chemotherapy with gemcitabine and docetaxel followed by concurrent radiation and continuous infusion 5FU and consolidation gemcitabine/docetaxel chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have biopsy-proven, resected with curative intent cholangiocarcinoma, gallbladder, pancreatic or ampullary adenocarcinoma.
* Patients must be 18 years or older.
* Patients must have a NCI CTC Performance Status of 0-2.
* Patients must not have any prior chemotherapy or radiation therapy for this current malignancy.
* At least 3 weeks should have elapsed since any surgery requiring general anesthesia.
* Patients must have no prior malignancies except for basal or squamous skin cancers, cervical carcinoma-in-situ, unless in remission for >5years
* Pregnant patients are not eligible. Non-pregnant status will be determined in all women of childbearing potential. All patients will be required to use an effective means of contraception if sexually active during therapy.
* Initial Required Laboratory Values:
* Absolute neutrophil count ≥ 1,500/mm3, platelet count ≥ 150, 000/mm3, and hemoglobin ≥ 9 g/dL.
* Serum creatinine should be ≤ 2 mg/dL.
* Serum bilirubin should be ≤ 3.0 mg/dL (biliary stents allowed).
* Serum transaminases should be ≤ 5-fold the institutional upper limits.
* Patients must not have any co-existing severe medical illnesses, such as unstable angina, uncontrolled diabetes mellitus, uncontrolled arrhythmia or uncontrolled infection.
* Patients must be able to sign an informed consent.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2002-09; Primary Completion 2010-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Tan, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participants enrollment on 09/14/2002 and closed to participant enrollment on 11/06/2012
Period: Overall Study
Arm/Group | Arm 1 (Gemcitabine, Docetaxel, 5FU, Radiation)
Started | 50
Completed | 48
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1 (Gemcitabine, Docetaxel, 5FU, Radiation)
Number analyzed (Participants) | 50
Age, Continuous [Median (Full Range); unit: years] | 59 [41 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 50
Overall stage [Number; unit: participants] — -There are some staging differences between biliary tract cancer, pancreatic cancer, and ampullary cancer but general staging information is listed below:
  * Stage I (best outcome) and Stage II means that there is only cancer in the primary site with no spread to local lymph nodes or spread to other sites of the body.
  * Stage III means that the cancer is in the primary site, possibly in nerves and blood vessels around the primary site, and may be in nearby lymph nodes.
  * Stage IV means that the cancer has spread to distant parts of the body (worst outcome)
  participants
    I | 3
    II | 46
    III | 1
    IV | 0
Disease type [Number; unit: participants]
  Pancreatic cancer | 29
  Biliary tract cancer | 12
  Ampullary cancer | 9
T-stage [Number; unit: participants] — * T describes the size of the main (primary) tumor and whether it has grown outside the primary site and into nearby organs.
  * T1 is generally associated with a better outcome and the outcome generally worsens as you increase the T number
  participants
    1 | 2
    2 | 11
    3 | 35
    4 | 2
N-stage [Number; unit: participants] — N describes the spread to nearby (regional) lymph nodes.
  X: Nearby (regional) lymph nodes cannot be assessed.
  N0: The cancer has not spread to nearby lymph nodes.
  N1: The cancer has spread to nearby lymph nodes.
  participants
    0 | 10
    1 | 36
    X | 4
Differentiation [Number; unit: participants] — Well-differentiated cancer cells look more like normal cells and tend to grow and spread more slowly than poorly differentiated or undifferentiated cancer cells.
  participants
    Well | 4
    Moderate | 17
    Poor | 28
    Not reported | 1
Lymphovascular involvement [Number; unit: participants]
  Yes | 36
  No | 9
  Not Reported | 5
CA 19-9 (tumor marker) [Number; unit: participants] — * Generally the higher the CA19-9 level the more the cancer is growing
  * High CA 19-9 levels can also be caused by non-cancerous conditions such as gallstones, a blockage of the bile duct (jaundice), pancreatitis, cystic fibrosis, and liver disease.
  participants
    <40 | 34
    40-100 | 11
    >100 | 5

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Severe Toxicities
Description: Toxicity was graded according to National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 2.0
Time Frame: 1 month after completion of treatment (treatment lasts approximately 19 weeks)
Measure: Number; unit: percentage of participants
Groups:
- Arm 1: Gemcitabine 1000 mg/m2 IV on Day 1 and Day 8 of a 21 day cycle for 2 cycles
  Docetaxel 35 mg/m2 IV on Day 1 and Day 8 of a 21 day cycle for 2 cycles
  5FU CIVI 225 mg/m2 per day throughout radiation (starts 3 weeks after start of cycle 2)
  Radiation 5040 cGy or 5400 cGy for positive margins (starts 3 weeks after start of cycle 2). Daily dose of 1.8 Gy five days per week.
  Gemcitabine 1000 mg/m2 IV on Days 1 and 8 of 21 day cycle for 2 cycles (this starts 4 weeks after radiation)
  Docetaxel 35 mg/m2 IV on Days 1 and 8 of 21 day cycle for 2 cycles (this starts 4 weeks after radiation)
Arm/Group | Arm 1
Number analyzed (Participants) | 48
percentage of participants | 20

2. Secondary Outcome: Toxicities Associated With Treatment (Grade 1-2)
Description: Toxicity was graded according to National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 2.0. The most common grade 1-2 non-hematologic and hematologic toxicities were collected for this outcome.
Time Frame: 30 days after completion of treatment (treatment lasts approximately 19 weeks)
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1
Number analyzed (Participants) | 48
percentage of participants
  Mucositis | 31
  Nausea | 48
  Vomiting | 23
  Diarrhea | 31
  Dehydration | 17
  Weight loss | 27
  Fatigue | 67
  Renal toxicity | 13
  Hepatotoxicity | 69
  Infection | 13
  Neutropenia | 46
  Anemia | 65
  Thrombocytopenia | 46

3. Secondary Outcome: Toxicities Associated With Treatment (Grade 3-4)
Description: Toxicity was graded according to National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 2.0. The most common grade 3-4 non-hematologic and hematologic toxicities were collected for this outcome.
Time Frame: 30 days after completion of treatment (treatment lasts approximately 19 weeks)
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1
Number analyzed (Participants) | 48
percentage of participants
  Mucositis | 2
  Nausea | 4
  Vomiting | 4
  Diarrhea | 15
  Dehydration | 4
  Weight loss | 0
  Fatigue | 8
  Renal toxicity | 0
  Hepatotoxicity | 4
  Infection | 15
  Neutropenia | 23
  Anemia | 4
  Thrombocytopenia | 6

4. Secondary Outcome: Disease Free Survival (DFS) - Median
Description: DFS was defined as the time from the initiation of treatment to relapse or death, whichever occurred first.
Time Frame: Median follow-up was 24 months (range 3.2-97 months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1
Number analyzed (Participants) | 48
months
  Pancreatic cancer | 9.6 [5.8 to 11.6]
  Biliary/ampullary cancer | 12.7 [7.9 to 18.9]

5. Secondary Outcome: Disease Free Survival (DFS) - Median
Description: DFS was defined as the time from the initiation of treatment to relapse or death, whichever occurred first.
Time Frame: Median follow-up was 24 months (range 3.2-97 months)
Population: 30 out of 48 participants completed all components of the study therapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1
Number analyzed (Participants) | 30
months
  Pancreatic cancer | 12.8 [5.9 to 17.5]
  Biliary cancer/ampullary cancer | 15.0 [8.1 to 18.9]

6. Secondary Outcome: Overall Survival (OS) - Median
Description: OS was defined as the time from the initiation of treatment to death from any cause or last follow-up.
Time Frame: Median follow-up was 24 months (range 3.2-97 months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1
Number analyzed (Participants) | 48
months
  Pancreatic cancer | 17.6 [8.6 to 23.8]
  Biliary cancer/ampullary cancer | 23.8 [11.4 to 47.0]

7. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the initiation of treatment to death from any cause or last follow-up
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1
Number analyzed (Participants) | 48
percentage of participants
  Pancreatic cancer | 60.7 [45.0 to 81.8]
  Biliary/ampullary cancer | 75.0 [58.0 to 96.6]

8. Post Hoc Outcome: Incidence of Disease Recurrence
Time Frame: Median follow-up was 24 months (range 3.2-97 months)
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1
Number analyzed (Participants) | 48
percentage of participants | 83

9. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the initiation of treatment to death from any cause or last follow-up
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1
Number analyzed (Participants) | 48
percentage of participants
  Pancreatic cancer | 32.1 [18.8 to 55.1]
  Biliary/ampullary cancer | 49.1 [31.2 to 77.3]

10. Secondary Outcome: Overall Survival (OS) - Median
Description: OS was defined as the time from the initiation of treatment to death from any cause or last follow-up.
Time Frame: Median follow-up was 24 months (range 3.2-97 months)
Population: 30 out of 48 participants completed all components of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1
Number analyzed (Participants) | 30
months
  Pancreatic cancer | 24.5 [9.7 to 29.4]
  Biliary cancer/ampullary cancer | 23.8 [12.8 to 70.4]

11. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the initiation of treatment to death from any cause or last follow-up
Time Frame: 1 year
Population: 30 out of 48 participants completed all components of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1
Number analyzed (Participants) | 30
percentage of participants
  Pancreatic cancer | 78.6 [59.0 to 100.0]
  Biliary/ampullary cancer | 81.2 [64.2 to 100.0]

ADVERSE EVENTS:
Arm/Group | Arm 1
Serious Adverse Events (participants affected / at risk) | 16/48
Other Adverse Events (participants affected / at risk) | 48/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=48)
Abdominal cystic lesion (Gastrointestinal disorders) | 1
Cavitary lung lesion (Respiratory, thoracic and mediastinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Death (General disorders) | 1
Dehydration (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Dizziness (Nervous system disorders) | 1
Edema (General disorders) | 1
Febrile neutropenia (Infections and infestations) | 1
Fever (General disorders) | 3
Generalized weakness (General disorders) | 1
Granulocytes (Investigations) | 1
Hemoglobin (Blood and lymphatic system disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
Ileus, GI (Gastrointestinal disorders) | 1
Infection (Infections and infestations) | 6
Leukopenia (Investigations) | 1
Nausea (Gastrointestinal disorders) | 1
Pain (General disorders) | 1
Platelets (Investigations) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Syncope (Nervous system disorders) | 1
Thrombosis/embolism (Vascular disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=48)
Alkaline phosphatase (Investigations) | 18
Alopecia (Skin and subcutaneous tissue disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 11
Anxiety (Psychiatric disorders) | 1
Ascites (Gastrointestinal disorders) | 2
BUN (Investigations) | 2
Bilirubin (Investigations) | 1
Chills (General disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Creatinine (Renal and urinary disorders) | 6
Dehydration (Gastrointestinal disorders) | 9
Depression (Psychiatric disorders) | 5
Diarrhea (Gastrointestinal disorders) | 21
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 1
Edema (General disorders) | 3
Erythema (Skin and subcutaneous tissue disorders) | 1
Eye (Eye disorders) | 1
Fatigue (General disorders) | 34
Fever (General disorders) | 2
Flatulence (Gastrointestinal disorders) | 1
Flushing (Vascular disorders) | 1
Granulocytes (Investigations) | 28
Hand/foot syndrome (Skin and subcutaneous tissue disorders) | 5
Hematochezia (Gastrointestinal disorders) | 1
Hematuria (Renal and urinary disorders) | 2
Hemoglobin (Blood and lymphatic system disorders) | 32
Hemorrhage (General disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 24
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypertension (Vascular disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 25
Hypocalcemia (Metabolism and nutrition disorders) | 16
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 9
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 9
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 3
Infection (Infections and infestations) | 7
Insomnia (Psychiatric disorders) | 4
Leukopenia (Investigations) | 32
Lymphopenia (Investigations) | 33
Mucositis (Gastrointestinal disorders) | 11
Nausea (Gastrointestinal disorders) | 23
Nocturia (Renal and urinary disorders) | 1
Other neurologic (Nervous system disorders) | 1
Pain (General disorders) | 25
Phlebitis (Vascular disorders) | 1
Platelets (Investigations) | 24
Proteinuria (Renal and urinary disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 2
SGOT/SGPT (Investigations) | 26
Sensory neuropathy (Nervous system disorders) | 2
Skin-photosensitivity (Skin and subcutaneous tissue disorders) | 1
Stomatitis (Gastrointestinal disorders) | 2
Sweating (General disorders) | 1
Thrombosis/embolism (Vascular disorders) | 2
Thrush (Infections and infestations) | 1
Urinary retention (Renal and urinary disorders) | 1
Urinary tract infection (Renal and urinary disorders) | 3
Vomiting (Gastrointestinal disorders) | 1
Weight loss (Gastrointestinal disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes